CLINICAL TRIAL: NCT03177421
Title: Improving Bedtime Media Use and Sleep Through Health Information Technology
Brief Title: Health Information Technology to Improve Bedtime Media Use in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study technology decommissioned at clinical site.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Randall Grout, Visiting Assistant Professor of Clinical Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: chsr_bedtime-media-cdss_2017
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Sleep Hygiene, Inadequate
MeSH Terms: conditions — Sleep Hygiene | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Midway through the study, participants from the control group will be folded into the intervention group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedtime media use and sleep problems (Experimental): This arm will receive screening for and associated clinical decision support on sleep problems and bedtime media use.
  Interventions: Other: Problematic bedtime media use counseling
- Sleep problems only (Other): This arm will receive screening for and associated clinical decision support on sleep problems only.
  Interventions: Other: Sleep problem counseling

INTERVENTIONS:
Other: Problematic bedtime media use counseling — Participants will be screened for bedtime media use and sleep problems, and the clinical decision support system will recommend counseling on the respective problems identified on screening.
  Other Names: Intervention
  Arms: Bedtime media use and sleep problems
Other: Sleep problem counseling — Participants will be screened for sleep problems, and the clinical decision support system will recommend counseling if problems are identified.
  Other Names: Control
  Arms: Sleep problems only

SUMMARY:
The objective of this study is to use health information technology to implement and evaluate a counseling recommendation for children who suffer from problematic sleep associated with bedtime media use. Participants will be randomized by clinic to be screened for basic sleep concerns and receive appropriate counseling, or to be screened for sleep concerns and media use, and receive appropriate counseling.

DETAILED DESCRIPTION:
Children and adolescents are increasingly integrating media and technology into daily life. A large body of research has shown poor sleep-related outcomes related to media exposure, especially in evening or bedtime hours - a trend that holds true from infancy to adolescence. Prior research has demonstrated clinic-based interventions can be effective in reducing general screen time. Yet, little work has been done to leverage existing health information technology to adapt bedtime media use guidelines into sustainable counseling interventions. This study will develop, implement, and evaluate a computerized, evidence-based decision support intervention for reducing inappropriate childhood bedtime media use and improving sleep measures.

ELIGIBILITY:
Inclusion Criteria:

* Attend a participating clinic
* Complete a prescreener form in the clinic

Exclusion Criteria:

* None

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60100 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Rate of clinician counseling for problematic bedtime media use and sleep problems | Up to 3 years

SECONDARY OUTCOMES:
Change in bedtime media use following clinician counseling | Up to 3 years
Change in inadequate sleep quantity following clinician counseling | Up to 3 years
Change in daytime sleepiness following clinician counseling | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall W. Grout, MD, MS, Principal Investigator — Indiana University - Ped Health Services
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No